CLINICAL TRIAL: NCT02815761
Title: A Prospective Study of Factors Related to Readmission and Mortality of COPD Patients in Hong Kong.
Brief Title: A Prospective Study Readmission and Mortality of COPD Patients
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fanny W.S. Ko, Honorary Associate Professor, Chinese University of Hong Kong
Other Study IDs: COPD readmssion_2011a
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be taken at first visit for assessment of inflammatory markers.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: NO intervention, just observation — No intervention.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common disease worldwide with a high burden on healthcare resources. The prevalence of COPD varied from 11.4 to 26.1% according to a recent multi-city population study using spirometry. In Hong Kong (HK), the prevalence rates of COPD in the elderly population aged ≥60 years were 25.9% and 12.4% based on the spirometric definition of forced expiratory volume in 1s (FEV1)/forced vital capacity (FVC) ratio <70% and the lower limit of normal of the FEV1/FVC respectively. In 2005, the crude mortality rate of COPD was 29.1/100 000, while the crude hospitalization rate was 193/100,000 in HK. In HK, COPD ranked second as a respiratory cause for hospitalization. In those 75 years or older, the hospitalization rate for COPD was as high as 2,225/100,000. The economic burden of COPD on the society is enormous.

Previous studies gave information on the overall morbidity, mortality and the prevalence of COPD in HK. One study compared the management of COPD patients in HK with other countries and found that COPD patients in HK were under-treated. No large scale study has looked into the details of COPD patients in HK, like their co-morbidities and how they are being treated and how these factors affect the readmission of these patients. Large prospective studies which incorporate all the potentially relevant variables are required to refine prediction of the important outcomes of AECOPD and thus to inform clinical decision making, for example on escalation of care, facilitated discharge and provision of palliative care.

DETAILED DESCRIPTION:
Aim of this study

The aim of this study is to assess the factors that are related to readmission and mortality of COPD patients in Hong Kong.

Method

This is a prospective observational study of patients. Patients who are admitted to the participating hospital with acute exacerbations of COPD (AECOPD) will be recruited. AECOPD was defined as occurring when a patient with background COPD11, with FEV1/FVC ratio <70%, presented with at least two major symptoms (increased dyspnea, increased sputum purulence, or increased sputum volume), or one major and one minor symptom (nasal discharge/congestion, wheeze, sore throat, or cough) for at least 2 consecutive days. Written informed consent will be obtained from each subject.

Inclusion criteria:

1. Subjects with a diagnosis of COPD according to the Global Initiative for chronic Obstructive Lung Disease (GOLD) Guideline16 with previous spirometry showing FEV1/FVC ratio of <0.70 with an AECOPD will be recruited for this study.
2. Age ≥40 years

Exclusion criteria:

1. Subjects who have been diagnosed with asthma, bronchiectasis or other chronic lung disease apart from COPD will be excluded
2. Patients with history of lung resection

4. Those who are unable to give consent Baseline assessments

1. Baseline assessments will be performed at 6-8 weeks after the AECOPD when the patients are at their stable state.
2. Demographic data including age, sex, body weight, height, smoking history, social history and medication usage, co-morbidities and any home oxygen or non-invasive positive pressure ventilation (NPPV) usage will be collected. Number of hospitalizations and accident and emergency department attendance in the past 12 month will be recorded. Any history of intubation or acute NPPV usage will be noted also.
3. American Thoracic Society (ATS) respiratory questionnaire17 will be asked.
4. Spirometry will be performed using the MICROLAB 3300 spirometer (Micro Medical, Kent, UK) in a sitting position, according to the ATS/European Respiratory Society (ERS) standards.18 Both pre- and post-bronchodilator (20 min after inhaling 400 mg of salbultamol [Ventolin; GlaxoSmithKline, E´ vreux, France] through a 500 mL spacer) tests will be performed. The updated predicted spirometric values for the Hong Kong Chinese were used.
5. Six min walk test will be performed according to the ATS guideline.
6. Modified Medical Research Council dyspnoea scale (MMRC)21 will be assessed.
7. St George's Respiratory Questionnaire (SGRQ)22 and medical outcomes short form 36 questionnaire (SF-36) 23 will be administered to all subjects.
8. Depression score
9. Blood saved for inflammatory markers analyses

Subsequent assessment:

Subjects will be reassessed every 12 months for repeat spirometry, 6 minute walk test, MMRC, SGRQ and SF-36 score for a total of 3 years. All hospitalizations, scheduled and unscheduled clinic visits in the subsequent 36 months after the baseline assessment will be recorded by asking the patient and with verification of their computer medical records. Any mortality (and the cause) will also be recorded.

Sample size:

This is a prospective observational study with primary aim to assess factors related to readmission and mortality of COPD patients in Hong Kong. We believe a sample size of 800 would be able to give us some meaningful data.

Data analysis:

Data will be analyzed by the Statistical Package of the Social Science (SPSS) Statistical software for Window, Version 17.0 (SPSS Inc, IL, USA). Descriptive statistics will be used and data will be presented as mean (SD) or median (IQR) as appropriate. Chi-square test, t-test, Mann-Whitney U test will be used to compare the clinical parameters of COPD patients with the different disease severities as appropriate. A p value of < 0.05 will be considered to be significant.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a diagnosis of COPD according to the Global Initiative for chronic Obstructive Lung Disease (GOLD) Guideline16 with previous spirometry showing FEV1/FVC ratio of <0.70 with an AECOPD will be recruited for this study.
2. Age ≥40 years

Exclusion Criteria:

1. Subjects who have been diagnosed with asthma, bronchiectasis or other chronic lung disease apart from COPD will be excluded
2. Patients with history of lung resection

4. Those who are unable to give consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study of patients. Patients who are admitted to the participating hospital with acute exacerbations of COPD (AECOPD) will be recruited. AECOPD was defined as occurring when a patient with background COPD11, with FEV1/FVC ratio <70%, presented with at least two major symptoms (increased dyspnea, increased sputum purulence, or increased sputum volume), or one major and one minor symptom (nasal discharge/congestion, wheeze, sore throat, or cough) for at least 2 consecutive days.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2013-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
COPD exacerbations | 3 years
  Exacerbations that required treatment with antibiotic or systemic steroid
Mortality | 3 years
  death

CONTACTS AND LOCATIONS:
Overall Officials: Fanny Ko, MD, Principal Investigator — fannyko@cuhk.edu.hk
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Ko FWS, Chan KP, Ngai J, Ng SS, Yip WH, Ip A, Chan TO, Hui DSC. Blood eosinophil count as a predictor of hospital length of stay in COPD exacerbations. Respirology. 2020 Mar;25(3):259-266. doi: 10.1111/resp.13660. Epub 2019 Aug 6. PMID 31385389